CLINICAL TRIAL: NCT02307201
Title: Magnesium Sulfate During the Postpartum in Women With Severe Preeclampsia Receiving Treatment for More Than 8 Hours Before Delivery. A Randomized Multicenter Clinical Trial .
Brief Title: Magnesium Sulfate During the Postpartum in Women With Severe Preeclampsia
Acronym: MAG-PIP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Complejo Hospitalario Dr. Arnulfo Arias Madrid (Other)
Responsible Party: Principal Investigator, Paulino Vigil-De Gracia, MEDICAL DOCTOR, GYNECOLOGY AND OBSTETRIC, Complejo Hospitalario Dr. Arnulfo Arias Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: complejoh
Record Dates: First submitted 2014-11-24; First posted 2014-12-04 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Post Partum Severe Preeclampsia
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Postpartum Magnesium sulfate (Experimental): The patient will receive magnesium sulfate as usual for 24 hours postpartum
  Interventions: Drug: Magnesium Sulfate
- No postpartum treatment (No Intervention): The patient did not receive postpartum magnesium sulfate or other anticonvulsant during 24 hours postpartum

INTERVENTIONS:
Drug: Magnesium Sulfate — The patient will receive magnesium sulfate for 24 hours postpartum
  Other Names: No postpartum treatment
  Arms: Postpartum Magnesium sulfate

SUMMARY:
There is no evidence that patients receiving magnesium sulfate before birth are required to maintain the drug for 24 hours. Therefore the investigators will have a randomized clinical study in patients with severe preeclampsia who have been treated with impregnation of magnesium sulphate and at least eight hours have received the drug before birth. If the patient agrees and signs the consent is randomized to: 1-receive sulfate for 24 hours postpartum as usual or, 2- not receiving the postpartum magnesium sulfate or other anticonvulsant drugs. This study can be conducted in 12 maternity latin america.

DETAILED DESCRIPTION:
The final treatment known for pre-eclampsia and eclampsia is the termination of pregnancy. However to prevent eclampsia in patients with severe pre-eclampsia has been demonstrated the effectiveness of magnesium sulfate. There are multiple studies that prove the effectiveness of magnesium sulfate to prevent eclampsia in patients with severe disorder of blood pressure during pregnancy. These studies used the drug before birth and continue after birth. Therefore the investigators can not conclude whether the administration just before pregnancy is sufficient to prevent seizure. If the cure or definitive treatment of pre-eclampsia is the interruption, did not seem necessary to justify the administration of drugs anti-eclampsia after birth. Obvious post delivery management with magnesium sulfate arises from the large number of postpartum eclampsia reported in many studies. It is unknown whether administration of magnesium sulfate for a minimum period before delivery, requires even keep the drug post partum.

In addition to magnesium sulfate postpartum, is necessary to maintain urinary catheter to monitoring the removal of magnesium sulfate; is usual to maintain the patient at all or almost all rest by monitoring sulfate and diuresis , this prevents a proper relationship mother and babe and even prevents breastfeeding during that period and is also known increased risk of secondary thromboembolism due to prolonged rest in the postpartum / caesarean section.Thus, maintain magnesium sulfate for 24 hours carries a higher cost, greater vigilance and some risks, without known real effect.

A randomized clinical study conducted by Belfort and colleagues and published in January 2003, where magnesium sulphate compared to nimodipine to prevent eclampsia in women with severe pre-eclampsia, showed interesting outcome. Such research analyzed 819 randomized patients in the nimodipine group and 831 in the magnesium sulfate group. Magnesium sulphate was better than Nimodipine in preventing eclampsia. Interestingly, the greater effectiveness of sulfate appears to prevent all eclampsia postpartum (9 vs 0) and obviously was used before the termination of pregnancy, however no difference compared with nimodipine in eclampsia before birth (12 vs 7).

There are two possible reasons for the non-appearance of postpartum eclampsia: 1- maintain postpartum magnesium sulfate, 2- dose 12-13 grams before birth disruption are sufficient to prevent eclampsia.

The MAGPIE study randomized 1335 postpartum patients (unused sulphate before delivery) using magnesium sulfate postpartum / cesarean (696 women) or placebo postpartum / cesarean (639 women), and found no significant difference in the amount of eclampsia . Thus, the use of magnesium sulfate for first time in the postpartum is not better to use a placebo. If the investigators combine the findings of eclampsia postpartum Belfort study and MAGPIE study is logical to think that the success of the Belfort study in the postpartum is not for the use of magnesium sulfate post delivery and not only due to the termination of pregnancy because there are postpartum eclampsia in the nimodipine group.

If the investigators consider unjustified use of magnesium sulfate postpartum, when maintained at least 8 hours before delivery, the investigators decided to make a non-inferiority randomized study.The investigators assume that using or not using magnesium sulfate during the postpartum prevents similar amount of postpartum eclampsia, if during pregnancy was used (impregnation and at least 8 hours before birth).

For all these reasons the investigators propose the following: A randomized trial is necessary where all those patients who received magnesium sulfate for at least 8 hours before birth (involves impregnation and maintenance 8 hours) will be randomized to two groups of study: 1- Continue magnesium sulfate for 24 hours and 2-not use magnesium sulfate or other anticonvulsant drug post delivery.

This study is planned in 12 maternity latin america

ELIGIBILITY:
Inclusion Criteria:

* Severe preeclampsia or severe preeclampsia aggregated to chronic hypertension with > 24 weeks of gestation treated with 4-6 grams of magnesium sulfate for impregnation with a minimum of 8 hours continuous of magnesium sulfate before delivery
* The study begins to terminate pregnancy

Exclusion Criteria:

* HELLP syndrome
* Eclampsia
* Renal insufficiency
* Diabetes mellitus
* Disease of collagen
* Heart disease

Ages: 14 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1114 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Eclampsia | 24 hours postpartum
  Convulsion after delivery in any group (with magnesium sulfate or without magnesium sulfate), during 24 hours postpartum.

SECONDARY OUTCOMES:
Postpartum hemorrhage | 24 hours postpartum
  Blood loss > 500 post vaginal delivery or > 800 cc post cesarean section, during 24 hours postpartum
Maternal respiratory distress | 24 hours postpartum
  clinical respiratory distress,during 24 hours postpartum
Grams of magnesium sulfate before delivery | 8 to 72 hours with magnesium sulfate before delivery
  Hours and grams of magnesium sulfate before delivery
Severe hypertension postpartum | 72 hours postdelivery
  Diastolic Blood pressure > 110 mmHg and/or systolic blood pressure > 160 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Paulino Vigil De Gracia, Principal Investigator — Complejo Hospitalario Dr. Arnulfo Arias Madrid; Jack Ludmir, MD, Study Chair — School of medicine, Pennsylvania Hospital. University de Pennsylvania. Philadelphia
Locations (9):
- Dominican Republic (2):
  - Hospital Materno Infantil san Lorezo de las Minas, Santo Domingo, Santo Domingo Province
  - Hospital Universitario Maternidad Nuestra señoa de Alta Gracia, Santo Domingo, Santo Domingo Province
- Hospital Teodoro Maldonado De Guayaquil, Guayaquil, Ecuador
- Hospital Primero de Mayo, San Salvador, El Salvador
- Panama (3):
  - Hospital Jose Domingo De Obaldia, Chiriquí, Chiriquí Province
  - Complejo Hospitalario Caja de Seguro Social, Panama City, Provincia de Panamá
  - Hospital Santo Tomás, Panama City, Provincia de Panamá
- Peru (2):
  - Hospital Regional de Cojamarca, Perú,, Cajamarca, Cajamarca Department
  - Instituto Materno perinatal, Maternidad de Lima, Lima, Lima Province

REFERENCES:
- [Background] Belfort MA, Anthony J, Saade GR, Allen JC Jr; Nimodipine Study Group. A comparison of magnesium sulfate and nimodipine for the prevention of eclampsia. N Engl J Med. 2003 Jan 23;348(4):304-11. doi: 10.1056/NEJMoa021180. PMID 12540643
- [Result] Altman D, Carroli G, Duley L, Farrell B, Moodley J, Neilson J, Smith D; Magpie Trial Collaboration Group. Do women with pre-eclampsia, and their babies, benefit from magnesium sulphate? The Magpie Trial: a randomised placebo-controlled trial. Lancet. 2002 Jun 1;359(9321):1877-90. doi: 10.1016/s0140-6736(02)08778-0. PMID 12057549